CLINICAL TRIAL: NCT01753895
Title: Comparison of Manual Blood Pressure Monitoring Using a Mercury Sphygmomanometer to an Automated Blood Pressure Instrument in a Research Setting
Brief Title: Mercury Versus Automated Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Arlene Hurley, Clinical Research Coordinator, Rockefeller University
Other Study IDs: AHU-0759
Record Dates: First submitted 2012-12-05; First posted 2012-12-20 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood pressure (BP) measurement is one of the most commonly performed screening tests in the clinical setting. Its accuracy is vital to the early diagnosis and effective management of hypertension, as emphasized by hypertension management guidelines. For most protocols being conducted in a clinical research setting, obtaining single or serial blood pressure reading(s) is often performed as a safety assessment, especially if the individual is participating in a study that requires a blood draw and/or the administration of a research drug, vaccine or device. It is imperative that the blood pressure data truly reflect the response, if any, the study participant experiences in relation to the research procedures and interventions.

DETAILED DESCRIPTION:
Despite the clear guidelines on manual blood pressure technique, there seems to be large inter-observer variations, both among nursing staff and physicians. These differences are further complicated by variables such as cuff selection and application, incorrect cuff positioning and rapid cuff deflation rate, inadequate rest period, and lack of repeated measurements. The blood pressure measurement obtained by an automated device is not as dependent on observer training and competency as the manual mercury device, yet its use requires careful patient evaluation for caffeine or nicotine use, cuff position, and proper wrist positioning, and instructing the individual not to move or talk if accurate blood pressures are to be obtained. If one performs the automated readings and manual blood pressure measurements under standardized conditions, the mean values will be quite similar; however, this possibility has not yet been fully tested.

Therefore, there is a need to assess systematically if there is in fact a difference in the two blood pressure monitoring approaches under controlled conditions. The goal of this study, then, is to examine our current practice of obtaining manual blood pressure measurement using a mercury sphygmomanometer compared to an automated wrist-mounted blood pressure device.

A possible implication of this study is if the blood pressure measurements using the automated blood pressure device are comparable to the measurements obtained using the mercury sphygmomanometer, than the mercury devices can be replaced by the more environmentally acceptable automated devices in our clinical research setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >18 and < 100 years of age
* With or without history of hypertension on or off antihypertensive medications
* Able to understand the information in the informed consent form and can provide written consent
* Upper arm and wrist access

Exclusion Criteria:

* Latex allergy
* Upper arm circumference > 52mm
* Wrist circumference < 5 inches and > 8 3/4 inches
* History of Mastectomy or Upper Extremity Peripheral Vascular Disease
* History of Carpal Tunnel Disease
* History of surgical repair of varicosities in the upper arm or wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assess difference in blood pressure readings in standard brachial vs. wrist-mounted radial blood pressure measurement | 1 outpatient visit and data will be analyzed at study completion
  This study will assess any differences in blood pressure readings noted between standard brachial blood pressure measurement and wrist-mounted radial blood pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Hurley, MA, ANP, CCRC, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States